CLINICAL TRIAL: NCT04922450
Title: A Multi-center, Single-arm, Phase II Clinical Study of Camrelizumab in Combination With Albumin Paclitaxel and Cisplatin for Neoadjuvant Treatment of Operable Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Clinical Study of Camrelizumab in Combination With Neoadjuvant Chemotherapy for Operable Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNIC21
Record Dates: First submitted 2021-05-24; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
Keywords: immunotherapy; PD-1 checkpoint inhibitor; neoadjuvant chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Immune Checkpoint Inhibitors; Cisplatin

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in our study.Participants will be given intravenous administration of Camrelizumab (200mg)，Albumin Paclitaxel(260mg/m²) and Cisplatin（80mg/m²）,After completing three times every three weeks of neoadjuvant therapy, The Participants will undergo surgery and Postoperative intensity modulated chemotherapy.Treatments will be administrated until death, or unacceptable toxicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab，albumin paclitaxel and cisplatin. (Experimental): Participants will be given intravenous administration of Camrelizumab (200mg)，Albumin Paclitaxel(260mg/m²) and Cisplatin（80mg/m²）,After completing three times every three weeks of neoadjuvant therapy, The Participants will undergo surgery and Postoperative intensity modulated chemotherapy. The duration of treatment will till death, or unacceptable toxicity show up.
  Interventions: Drug: PD-1 inhibitor; Drug: Albumin Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: PD-1 inhibitor — Intravenous administration of SHR1210 (200mg/3weeks)
Drug: Albumin Paclitaxel — Albumin Paclitaxel(260mg/m²),every 3 weeks
Drug: Cisplatin — Cisplatin（80mg/m²）, every 3 weeks

SUMMARY:
In this single-arm study, pathologically confirmed advanced head and neck squamous cell carcinoma will be enrolled to investigate the efficacy and safety of Camrelizumab in combination With albumin paclitaxel and cisplatin.

DETAILED DESCRIPTION:
First, the patient received neoadjuvant therapy once every three weeks for a total of three cycles（Camrelizumab in combination With albumin paclitaxel and cisplatin）.After the neoadjuvant treatment, the patient undergoes surgery and postoperative radiotherapy.According to the surgical margin and postoperative pathological conditions, combined with cisplatin concurrent chemotherapy as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years, both men and women;
2. Patients who diagnosed as Squamous cell carcinoma by pathological examination;
3. Patients who have not received systemic or local treatment for head and neck squamous cell carcinoma;
4. The primary tumor and lymph nodes can be completely surgically removed;
5. Exclude distant metastasis through chest CT and full-body bone scanning;
6. The patient's vital organs are functioning normally and can tolerate the specified treatment plan Absolute neutrophil count ≥1.8 × 109 / L platelets ≥100 × 109/L, Hemoglobin ≥9g/dL, serum albumin ≥3g/dL Bilirubin≤1.5 ULN ALT and AST≤2.5 ULN INR≤1.5 ULN leukocyte≥2000/L Serum creatinine ≤ 1.5 ULN Thyroid Stimulating Hormone≤ 1 ULN
7. ECOG score：0-1
8. Women of childbearing age (15-49 years old) have a negative serum or urine HCG test within 7 days before treatment, and agree to use medically approved measures for contraception during treatment and 120 days after treatment ends
9. Males who have not been sterilized must agree to take effective contraceptive measures during the study period and at least 120 days after the last dose of PD-1 monoclonal antibody
10. Patients can provide enough tissue samples for PD-L1 detection or exploratory research.
11. The patient signs an informed consent and voluntarily participates in the clinical trial

Exclusion Criteria:

1. Patients who pathologically confirmed non-squamous cell carcinoma
2. Patients who has recurrence or distant metastasis
3. Local lesions have been surgically removed
4. Patients who have received systemic anti-cancer therapy, including hormone therapy
5. Patients who have received treatment targeting PD-1 or PD-L1
6. Patients with active autoimmune disease or a history of autoimmune disease but may relapse(Patients with the following diseases are not excluded and can be further filtered)

   1. Controlled type 1 diabetes
   2. Hypothyroidism(If it can be controlled with hormone replacement therapy)
   3. Controlled celiac disease
   4. Skin diseases that do not require systemic treatment such as Vitiligo, Psoriasis and Hair loss.
   5. Any other disease that is not expected to recur without external triggers
7. Any active malignant tumors within 2 years before treatment, except for the specific cancers being studied in this trial and locally recurring cancers that have been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical in situ Cancer or breast cancer)
8. Any disease requiring systemic treatment with corticosteroids (referring to treatment with a dose higher than 10 mg/day of prednisone or equivalent doses of similar drugs) or other immunosuppressive treatments within 14 days before treatment.

   However, patients who have currently or previously used any of the following steroid regimens can be selected:
   1. Adrenaline replacement steroids(Prednisone ≤10mg/day or equivalent dose of similar drugs)
   2. Local, ophthalmic, intra-articular, intranasal and inhaled corticosteroids which is Systemic absorbed Minimally
   3. Prophylactically short-term (≤7 days) use of corticosteroids (for example, allergy to contrast agents) or for the treatment of non-autoimmune conditions (for example, delayed hypersensitivity reactions caused by contact allergens)
9. Uncontrolled diabetes within 14 days before treatment or laboratory abnormalities with potassium, sodium and corrected calcium levels> 1 after standard drug treatment or hypoalbuminemia grade ≥ 3
10. History of the following diseases: interstitial lung disease, non-infectious pneumonia or uncontrollable diseases, including pulmonary fibrosis, acute lung disease, etc.
11. Severe chronic or active infection (including tuberculosis infection, etc.) that required systemic antibiotics, antibacterial or antiviral treatment occurred within 14 days before the first administration of the study drug
12. The patient is known to have been infected with HIV
13. Untreated patients with chronic hepatitis B or HBV carriers with chronic hepatitis B virus (HBV) DNA ≥ 500 IU/mL or active hepatitis C virus carriers (HCV) should be excluded.

    Patients can be selected who is Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA <500 IU/mL) and cured hepatitis C patients.
14. Any surgery requiring general anesthesia has been performed within 28 days before treatment
15. Have had allogeneic stem cell transplantation or organ transplantation
16. Have any of the following cardiovascular risk factors:

    1. Cardiogenic chest pain within 28 days before treatment(moderate pain that restricts instrumental activities of daily living)
    2. Symptomatic pulmonary embolism within 28 days before treatment
    3. Acute myocardial infarction within 6 months before treatment
    4. Any history of heart failure that has reached Grade III or IV as defined by the New York Heart Association within 6 months before treatment
    5. Grade 2 ventricular arrhythmia within 6 months before the first administration of the study drug
    6. Have a history of cerebrovascular accident within 6 months before the first administration of the study drug
17. Have a history of severe hypersensitivity to other monoclonal antibodies
18. Patients with treatment toxicity (caused by previous anti-cancer treatments) have not returned to baseline or stabilized, unless it is an AE that is not considered a possible safety risk (such as hair loss, neuropathy, or specific laboratory abnormalities)
19. History of allergic reactions to cisplatin or other platinum-containing compounds
20. Peripheral nerve disease ≥ Grade 2 defined by NCI CTCAE v5.0 standard Have gotten a live vaccine within 4 weeks before treatment(Seasonal flu vaccines are usually inactivated vaccines and are allowed to be used; The vaccine used in the nasal cavity is a live vaccine and is not allowed to be used)
21. Abuse or dependence on alcohol or drugs and Basic medical conditions (including laboratory abnormalities) that are not conducive to the administration of the study drug , affect the interpretation of drug toxicity or AEs, lead to insufficient compliance with the study execution and possible damage
22. The patient participates in another therapeutic clinical study at the same time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate(CRR) | immediately after the surgery
  the short-term efficacy of Camrelizumab combined with albumin paclitaxel/cisplatin neoadjuvant treatment of operable locally advanced head and neck cancer
Pathological remission rate(PRR) | immediately after the surgery
  the short-term efficacy of Camrelizumab combined with albumin paclitaxel/cisplatin neoadjuvant treatment of operable locally advanced head and neck cancer

SECONDARY OUTCOMES:
2-year survival rate, 2-year progression-free survival rate, 2-year recurrence-free survival rate, 2-year survival rate without distant metastasis | 2 year
  1. the long-term efficacy of Camrelizumab combined with albumin paclitaxel/cisplatin neoadjuvant treatment of operable locally advanced head and neck cancer
Adverse event rate | 2 year
  The safety of Camrelizumab combined with albumin paclitaxel/cisplatin neoadjuvant treatment of operable locally advanced head and neck cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yaqian Han, Principal Investigator — Hunan Cancer Hospital; Wenxiao Huang, Principal Investigator — Hunan Cancer Hospital; Hui Wang, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author of published work.